CLINICAL TRIAL: NCT00385866
Title: Addressing Disparities in Cancer Care for Latino Medicare Beneficiaries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0120060236
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Cancer
Keywords: Patient Navigator; Community health; Communication
MeSH Terms: conditions — Neoplasms; Communication | interventions — Mass Screening; Patient Navigation; Educational Status

ARMS (2):
- Comparison Group (Active Comparator): The control or lesser intervention group, will receive cancer screening information on a quarterly basis, with no facilitation of services.
  Interventions: Behavioral: cancer screening and health education
- Intervention group (Active Comparator): The intervention group are those participants who were randomly assigned to receive facilitation of services in the form of patient navigation for the duration of the study.
  Interventions: Behavioral: cancer screening and health education; Behavioral: facilitation of Services to improve cancer screening

INTERVENTIONS:
Behavioral: cancer screening and health education — The control group will receive cancer screening and health education materials on a quarterly basis but will not have access to patient navigation services.
  Other Names: patient navigation; cancer screening and education
Behavioral: facilitation of Services to improve cancer screening — The intervention group will receive cancer education and faciliation of services in the form of patient navigation
  Other Names: patient navigation; faciliation of services; screening
  Arms: Intervention group

SUMMARY:
To reduce Cancer health care disparities that exists among minority Medicare beneficiaries and to demonstrate cost effectiveness of patient navigation in reducing the burden of cancer.

DETAILED DESCRIPTION:
The Latino population is the fastest growing minority population in the United States . Cancer ranks as the second leading cause of death among Latinos in the United States (24%), second only to heart disease . This project will evaluate whether an innovative facilitation program (targeting cancers of the prostate, colon/rectum, breast, and cervix) will improve cancer outcomes among Latino Medicare beneficiaries in the city of Newark, New Jersey.

The overall aim of this project is to institute an innovative cancer care facilitation program for elderly Latinos in the city of Newark, NJ. The goal is to reduce the disparities observed in screening, time to diagnosis and treatment services, by utilizing a multidisciplinary team approach to health care, incorporating systems thinking methodology. Using the Multilevel Approach to Community Health (MATCH) planning model , the program will incorporate community outreach, education, and access to screening, and patient assistance in all aspects of the health care continuum. It will also include cultural and linguistic competency training for all those involved in the facilitation process. To accomplish this goal, we propose four objectives:

1. To establish a multidisciplinary team that will utilize a systems thinking approach to design and structure the delivery of cancer screening, diagnosis and treatment facilitation services.
2. To build a collaborative consortium between program partners to improve screening outcomes, that will encourage the utilization of services in the community.
3. To improve the delivery of cancer prevention and treatment facilitation by providing cultural and linguistic competency training to the multidisciplinary team, providers, and the community.
4. To demonstrate the effectiveness of the intervention in reducing the burden of cancer, by increasing screening rates, improving time to diagnosis and delivery of treatment services, patient satisfaction, and appropriate use of Medicare services.

ELIGIBILITY:
Inclusion Criteria:

Cancer-Negative Group

1. Be of Hispanic/Latino Origin
2. Fluent in English and/or Spanish
3. Recipient of, Medicare Part A & B, or combined Medicare/Medicaid
4. Not having a previous diagnosis of cancer
5. Be capable of giving written informed consent prior to any study related procedures.
6. Be available and willing to complete all study assessments as specified.

Cancer-Positive Group

1. Be of Hispanic/Latino Origin
2. Fluent in English and/or Spanish
3. Recipient of, Medicare Part A & B, or combined Medicare/Medicaid
4. Having a previous diagnosis of cancer of the breast, cervix, colon and/or rectum, prostate, or lung.
5. Be capable of giving written informed consent prior to any study related procedures.
6. Be available and willing to complete all study assessments as specified.

Exclusion Criteria:

1. Member of the Medicare Advantage Plan, any Medicare managed care plan (Those who join the Medicare Advantage plan or a managed care plan during the course of the study will become ineligible to continue.)
2. Medicaid only beneficiaries
3. Institutionalized
4. Unable to provide written informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1272 (Actual)
Dates: Start 2006-10; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Reduce the disparities observed in utilization of cancer screening services | 2-4 years

SECONDARY OUTCOMES:
Improve the time to diagnosis and treatment services (resulting in reduced cost of cancer care | 4 years
Improve patient satisfaction and informed decision making. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ana Natale-Pereira, MD, MPH, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ, Newark, New Jersey, United States